CLINICAL TRIAL: NCT05217459
Title: A Prospective, Multicenter, Objective Performance Criteria Study to Evaluate the Efficacy and Safety of an Intracranial Self-expanding Drug Eluting Stent System for Symptomatic Intracranial Atherosclerotic Disease
Brief Title: The Efficacy and Safety of Intracranial Self-expanding DES in Symptomatic Intracranial Atherosclerotic Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sinomed Neurovita Technology Inc. (Industry)
Collaborators: Changhai Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNSC-202103
Record Dates: First submitted 2022-01-04; First posted 2022-02-01 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2024-05

CONDITIONS: Intracranial Arterial Diseases; Stent Restenosis; Percutaneous Transluminal Angioplasty
Keywords: Self-expanding intracranial stent; Symptomatic Intracranial Atherosclerotic Disease; In-stent restenosis
MeSH Terms: conditions — Intracranial Arterial Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Self-expanding intracranial drug stent system (Experimental): All patients receive Percutaneous transluminal angioplasty and stenting with self-expanding intracranial drug stent system (Temporary abbreviations: SINOMED IS-DES)
  Interventions: Device: Self-expanding intracranial drug stent system

INTERVENTIONS:
Device: Self-expanding intracranial drug stent system — All patients receive Percutaneous transluminal angioplasty and stenting with self-expanding intracranial drug stent system (Temporary abbreviations: SINOMED IS-DES)

SUMMARY:
The primary objective of this trial is to evaluate the safety and efficacy of SINOMED IS- DES in patients with symptomatic intracranial atherosclerotic stenosis.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, objective performance criteria clinical trial to evaluate the safety and efficacy of intracranial self-expanding drug stent system in the treatment of symptomatic intracranial atherosclerotic stenosis. A total of 128 patients are planned to be included. The primary endpoint is the incidence of In-stent restenosis at 6 months after operation (ISR is defined as stenosis greater than 50% within or immediately adjacent (within 5 mm) to the implanted stents and absolute luminal loss greater than 20% at 6 months follow-up imaging.). All patients will have clinical follow-up during intraoperative, 30 days, 6 months, 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. 30 to 75 years of age;
2. Patients with symptomatic intracranial atherosclerotic stenosis who failed antiplatelet therapy or poor collateral circulation compensation or hypoperfusion in the territory of the culprit artery;
3. Digital Subtraction Angiography(DSA) showed 70% to 99% stenosis in target intracranial artery
4. The target lesion was in the internal carotid artery (intracranial segment), middle cerebral artery, vertebral artery (intracranial segment), basilar artery, and it was a single lesion that required surgical treatment;
5. The target lesion reference diameter must be visually estimated to be ≥2.0 mm and <4.5mm in diameter, and lesion length of ≤34 mm;
6. mRS < 3;
7. The onset of the latest transient ischemic attack (TIA) was not limited or ischemic stroke occurred within 2 weeks prior to stenting procedure;
8. Willingness to participate in this clinical trial and signing the consent form, and be able to complete the corresponding inspections, follow-ups, etc. according to the requirements of the clinical protocol during the clinical trial.

Exclusion Criteria:

1. The target vessels was complete occlusion;
2. >70% stenosis observed at the intracranial large-vessel distal to the target vessel or >70% stenosis observed at the intracranial/extracranial large-vessel proximal to the target vessel;
3. Preoperative magnetic resonance only showed perforating infarction in the target lesion area;
4. Preoperative CT or MRI showed that there was hemorrhage transformation after infarction in the target vessel area, or a history of primary cerebral hemorrhage, or a history of subarachnoid, subdural and epidural hemorrhage within 30 days before operation, or there was no treatment Chronic subdural hematoma ≥5mm;
5. Hospitalized surgical treatment within 30 days before operation, or planned hospitalized surgical treatment within 6 months after surgery;
6. CT showed Severe calcified lesions;
7. Previously received endovascular treatment or surgical intervention at the target vessel (except for patients with simple balloon dilatation);
8. Non-atherosclerosis lesions;
9. Patients with potential sources of cardiac embolism (such as atrial fibrillation, left ventricular thrombosis, myocardial infarction within 6 weeks);
10. Concomitant intracranial tumor, aneurysm or intracranial arteriovenous malformation;
11. Known hypersensitivity to aspirin, heparin, clopidogrel, rapamycin (sirolimus), lactic acid polymer, poly-n-butyl methacrylate, nickel-titanium alloy, or contraindications to anesthetics and contrast agents;
12. Hemoglobin <100g/L, platelet count <100*109/L, International normalized ratio (INR) >1.5 (irreversible) or uncorrectable hemorrhagic factors;
13. Uncontrollable severe hypertension (systolic blood pressure>180mmHg or diastolic blood pressure>110mmHg)；
14. Known liver or renal insufficiency (ALT> 3x upper limit or AST > 3x upper limit, Serum creatinine>250μmol/L);
15. Life expectancy < 1 year;
16. Pregnant/lactating female patients;
17. Patients with cognitive impairment or mental diseases (except for those with cognitive impairment due to arterial stenosis);
18. Patients who were participated in other clinical trials within 3 months or participating in other clinical trials who had not yet reached the primary clinical endpoint;
19. Inapplicable for intravascular stenting treatment as per investigators judgment.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
The incidence of In-stent restenosis within 6 months after operation | 6 months after operation
  ISR is defined as stenosis greater than 50% within or immediately adjacent (within 5 mm) to the implanted stents and absolute luminal loss greater than 20% at 6 months follow-up imaging.

SECONDARY OUTCOMES:
Stent success | Immediately after operative
  Stent success is defined as ISS is successfully implanted into the vascular site of the target lesion with balloon pretreatment and the delivery system was successfully withdrawn.
Procedure success | Immediately after operative
  Procedure success is defined as a reduction in the degree of stenosis to ≤ 30% after the application of any interventional treatment method.
Percent of Participants With National Institutes of Health Stroke Scale (NIHSS) Score = 0 or 1 at 6 months follow-up | 6 months after operation
  The National Institutes of Health Stroke Scale (NIHSS) is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. A trained observer rates the patent's ability to answer questions and perform activities. Ratings for each item are scored with 3 to 5 grades with 0 as normal, and there is an allowance for untestable items. The range of scores is from 0 (normal) to 42 (profound effect of stroke on patient).
Rate of good functional outcomes measured by Modified Rankin Score (mRS) | 30days, 6 months, 1 year after operation
  Modified rankin score measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The range is 0-6 (0 is highest function with no symptoms and 6 is death). This outcome measured percentage of subjects with a "good" functional outcome with a score ranging from 0-2.
Rate of all revascularization and target lesion revascularization | 30days, 31days to 6 months, 1 year after operation
  The proportion of patients who had revascularization in target lesion or not
Symptomatic ISR within 6 months | within 6 months
  Symptomatic ISR is defined as ISR associated with ischemic event in the territory
Any stroke or death within 30 days after operation, and the incidence of recurrent ischemic stroke in the target vascular area within 31 days to 6 months, 1 year after operation. | 30days, 31days to 6 months, 1 year after operation
  As a composite endpoint include any stroke or death within 30 days, and the incidence of recurrent ischemic stroke in the target vascular area within 31 days to 6 months, 1 year after operation.
Any stroke or death within 30 days after operation | Within 30 days after operation
  Any stroke, death means death from any cause, including stroke or cerebrovascular disease
Stroke (including hemorrhage or ischemic stroke) or death within 30 days associated with the target vessel | Within 30 days after operation
  The proportion of patients who had any stroke or died within 30 days after operation in association with stenting implantion
The incidence of recurrent ischemic stroke in the target vascular area within 31 days to 6 months, 1 year after operation. | 31days to 6 months, 1 year after operation
  There is clear imaging evidence to confirm that the target vessel area is occluded again, which leads to ischemic stroke.
The incidence of recurrent ischemic stroke outside the target vascular area within 31 days to 6 months, 1 year after operation. | 31 days to 6 months, 1 year after operation
  There is clear imaging evidence to confirm that outside the target vessel area is occluded again, which leads to ischemic stroke.
Any parenchymal hemorrhage, subarachnoid hemorrhage or intraventricular hemorrhage | 31 days to 6 months, 1 year after operation
  There is clear imaging evidence to confirm that the incidence of any parenchymal hemorrhage, subarachnoid hemorrhage or intraventricular hemorrhage
All cause death | 31days to 6 months, 1 year after operation
  The proportion of patients who died from all causes is evaluated from 31 days to 6 months, 1 year after operation
Adverse events or severe adverse event | 31 days to 6 months, 1 year after operation
  The proportion of Adverse events or severe adverse event
Incidence of device defects | During operation
  The proportion of device defects in the process of testing, such as label errors, quality problems, malfunctions, etc.

CONTACTS AND LOCATIONS:
Overall Officials: jianming Liu, M.D/Ph.D, Principal Investigator — Changhai Hospital
Locations (14):
- China (14):
  - Beijing Chao-Yang Hospital, Capital Medical University, Beijing
  - The First Hospital of Jilin University, Changchun
  - The First People's Hospital of Changzhou, Changzhou
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Hangzhou First people's Hospital, Zhejiang University School of Medicine, Hangzhou
  - The First Affiliated Hospital of Harbin Medical University, Ha’erbin
  - The First Affiliated Hospital of USTC Anhui provincial hospital, Hefei
  - Qilu Hospital, Shandong University, Jinan
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Changhai Hospital, Shanghai
  - Shanghai Fourth People's Hospital, Shanghai
  - The First Hospital of Hebei Medical University, Shijiazhuang
  - Yantai Yu Huang Ding hospital, Yantai
  - The First Affiliated hospital of Zhengzhou hospital, Zhengzhou